CLINICAL TRIAL: NCT03001440
Title: Subject Understanding of the Risks Associated With ZYBAN®, WELLBUTRIN®, WELLBUTRIN SR®, and WELLBUTRIN XL®
Brief Title: A 7-year Assessment on Subject Understanding of ZYBAN/ WELLBUTRIN Associated Risks
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Collaborators: United Biosource Corporation (UBC) (Unknown)
Responsible Party: Sponsor
Other Study IDs: 205913
Record Dates: First submitted 2016-12-20; First posted 2016-12-23 (Estimated); Last update posted 2018-02-13 (Actual); Status verified 2018-02

CONDITIONS: Depressive Disorder, Major
Keywords: REMS; Smoking cessation; WELLBUTRIN; ZYBAN; Neuropsychiatric adverse events
MeSH Terms: conditions — Depressive Disorder, Major; Smoking Cessation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ZYBAN/WELLBUTRIN users: Subjects who currently use or who have filled a prescription for ZYBAN, WELLBUTRIN, WELLBUTRIN SR, or WELLBUTRIN XL for smoking cessation within the previous 6 months will be included in the study. Subjects will be required to complete the KAB survey either online or through a telephone interview.
  Interventions: Other: KAB survey

INTERVENTIONS:
Other: KAB survey — The KAB survey will be conducted among study population to evaluate their understanding of the potential serious risk with the use of ZYBAN. The 20 minutes survey can be completed either online or through a telephone interview.

SUMMARY:
Branded bupropion hydrochloride products including ZYBAN and WELLBUTRIN range are approved for the treatment of smoking cessation and depressive disorders respectively. The Risk Evaluation and Mitigation Strategy (REMS) for ZYBAN was initially approved in 2010 and consists of a Medication Guide and a timetable for REMS assessments submission at 18 months, 3 years and 7 years from the date of initial approval of REMS. The present study is a 7-year REMS assessment to evaluate subjects' understanding of the potential serious risk of neuropsychiatric adverse events associated with the use of ZYBAN, WELLBUTRIN, WELLBUTRIN SR, and WELLBUTRIN XL. The assessment will be a 20-minutes Knowledge, Attitudes and Behavior (KAB) survey and will be conducted among approximately 125 subjects currently using or who have filled a prescription for a branded bupropion product for smoking cessation within the 6 months prior to survey administration. ZYBAN, WELLBUTRIN, WELLBUTRIN SR, and WELLBUTRIN XL are registered trade marks of the GSK group of companies.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who currently use or who have filled a prescription for ZYBAN, WELLBUTRIN, WELLBUTRIN SR, or WELLBUTRIN XL for smoking cessation within the previous 6 months. (Note: Branded bupropion hydrochloride product use will be confirmed through a series of questions within the screener concerning manufacturer information detailed on the product label [label on medication container] and following a review of photographs of generic bupropion, ZYBAN, WELLBUTRIN, WELLBUTRIN SR or WELLBUTRIN XL tablet types online or via a paper copy sent with the invitation letter for those who choose to participate via phone)
* 18 years of age or older
* Fluent English speaker (for telephone)
* Consent to take the online survey or have the survey administered via a telephone interview

Exclusion Criteria:

* Subjects taking generic bupropion
* Subjects who currently use or who have filled a prescription for a branded bupropion product for depression alone
* Under 18 years of age
* Previous participation in a branded bupropion hydrochloride survey, which will be determined via self-report in the survey

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects of age 18 years or older who are currently using or who have filled a prescription for branded bupropion hydrochloride products including ZYBAN, WELLBUTRIN, WELLBUTRIN SR, WELLBUTRIN XL within the 6 months prior to survey administration for smoking cessation.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2016-10-07 (Actual); Primary Completion 2016-12-28 (Actual); Study Completion 2016-12-28 (Actual)

PRIMARY OUTCOMES:
Number (No.) of subjects correctly responding to individual survey questions | 7 years
  The proportion of correct answers to survey questions concerning the risks associated with branded bupropion hydrochloride products will be summarized by use of formulation of ZYBAN or WELLBUTRIN. Smoking behavior, demographic information, information related to the receipt and reading of the Medication Guides and how the branded bupropion hydrochloride product is normally received will also be reported. Point estimates for the proportion with correct responses will be calculated for each question about the risks of branded bupropion products. In the case of multiple choice questions, the number and proportion of subjects reporting each response will also be provided.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline